CLINICAL TRIAL: NCT02902367
Title: Effects of Sms-guided Outdoor Walking and Strength Training After Acute Stroke and TIA - a Randomized Controlled Trial
Brief Title: Sms-guided Training After Acute Stroke or Transient Ischemic Attack - a Randomized Controlled Trial
Acronym: SMS/TIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Birgit Vahlberg, Md Dr, RPT, Uppsala County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UppsalaCC2
Record Dates: First submitted 2016-09-11; First posted 2016-09-15 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Acute Stroke; TIA (Transient Ischemic Attack)
Keywords: mobility; exercise; walking capacity; fat mass; muscles
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Motor Activity | interventions — Exercise; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: (Experimental): Outdoor walking and strength exercise, Three months, daily SMS.
  Interventions: Other: Outdoor walking and strength exercise
- Control group (Other): Usual care; no restriction for exercise, Three months
  Interventions: Other: control group

INTERVENTIONS:
Other: Outdoor walking and strength exercise — Exercise group: Participants are supposed to perform an outdoor walking exercise program and one strength exercise for 12 weeks. The first 2 weeks start with daily walks. The intensity and frequency of walks will progressively increase performed according to the Borg scale: 12-15, ie, moderate to strenuous. Participants will walk 5-7 days/week. Added to this is a strength exercise, i.e. chair-rising which also should be performed daily.
  Other Names: exercise
  Arms: Intervention:
Other: control group — Control-Group: Treatment as usual for 12 weeks, without restriction of being physically active.
  Other Names: control
  Arms: Control group

SUMMARY:
Eighty community-living individuals in Uppsala municipality will be included. Intervention: Outdoor walking exercise program and one strength exercise. Methods: Clinical assessments, questionnaires and medical records. Assessment of motor function, cognition, level of physical activity, food intake and perceived stress are performed at screening as baseline measurements. Walking capacity, mobility, handgrip strength, body composition and cardiovascular risk markers will be assessed at baseline and after 12 week of training. At one year after training health-related quality of life, another cardiovascular incidence and mortality will be documented.

DETAILED DESCRIPTION:
Eighty community-living individuals in Uppsala municipality will be included in a randomized controlled trial with two arms.

Intervention: Participants will perform an outdoor walking exercise program together with one strength exercise for 12 weeks. The intensity and frequency of the training will progressively increase. Participants are supposed to walk and perform strength training 5-7 days/week.

Methods: Clinical assessments, questionnaires and medical records used for documentation of age, sex, comorbidity, blood pressure, medications and previous education.

Assessment of motor function, cognition, level of physical activity, food intake and perceived stress are performed at screening as baseline measurements. Walking capacity (primary outcome measure), mobility, handgrip strength, body composition and cardiovascular risk markers will be assessed at baseline and after 12 week of training. At one year after training health-related quality of life, another cardiovascular incidence and mortality will be evaluated.

Power analysis is performed. The investigators will analyze the data using an intention-to -treat analysis. Participants should have participated in at least 50% of the training sessions

ELIGIBILITY:
Inclusion Criteria:

1. Verified ischemic cerebral infarction or intracerebral hemorrhage.
2. Sufficient walking capacity and motor function
3. Able to communicate in Swedish
4. Signed consent

Exclusion Criteria:

One or more of the following:

1. Subarachnoid bleeding
2. Insufficient cognition and impaired ability to understand instructions
3. Medical problems that make it unsuitable to participate
4. Pacemaker (body composition measurements)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-03 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test (6MWT) | from baseline walking capacity to three months
  walking capacity

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | from baseline SPPB to three months
  mobility
10 meter walk test (10mWT) | from baseline 10mWT to three months
  gait speed
Hand-dynamometer (Jamar) | from baseline Jamar to three months
  hand-grip strength
Body composition (bioelectric impedance analysis) | from baseline body composition to three months
  muscles and fat mass and BMI
Cardiometabolic risk markers | from baseline cardiometabolic risk markers to three months
  blood lipids, c-reactive proteins (CRP), blood glukos, HbA1c, Insulin-like growth factor (IGF-1), Interleukin-6 (Il-6)
Heart and lung foundation stress test | at baseline
  self-perceived stress
Food frequency questionnaire | at baseline
  self-reported food intake and quality
Montreal outcome assessment (MoCA) | at baseline
  cognition
Modified rankin scale (MRS) | at baseline
  motor function
Mortality | from baseline to 1 year
  register-based mortality
Health-related quality of life | from baseline to 1 year
  register-based quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Vahlberg, Principal Investigator — Sweden,Uppsala Uppsala University Hospital
Locations (1):
- Birgit Vahlberg, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vahlberg BM, Eriksson S, Holmback U, Lundstrom E. Factors associated with changes in walking performance in individuals 3 months after stroke or TIA: secondary analyses from a randomised controlled trial of SMS-delivered training instructions in Sweden. BMJ Open. 2024 Mar 4;14(3):e078180. doi: 10.1136/bmjopen-2023-078180. PMID 38443081
- [Derived] Vahlberg BM, Lundstrom E, Eriksson S, Holmback U, Cederholm T. Potential effects on cardiometabolic risk factors and body composition by short message service (SMS)-guided training after recent minor stroke or transient ischaemic attack: post hoc analyses of the STROKEWALK randomised controlled trial. BMJ Open. 2021 Oct 18;11(10):e054851. doi: 10.1136/bmjopen-2021-054851. PMID 34663672
- [Derived] Vahlberg B, Lundstrom E, Eriksson S, Holmback U, Cederholm T. Effects on walking performance and lower body strength by short message service guided training after stroke or transient ischemic attack (The STROKEWALK Study): a randomized controlled trial. Clin Rehabil. 2021 Feb;35(2):276-287. doi: 10.1177/0269215520954346. Epub 2020 Sep 18. PMID 32942914